CLINICAL TRIAL: NCT01417767
Title: Phase 2/3 Study of Efficacy Study of CHG Regimen vs Decitabine to Treat Higher-risk MDS
Brief Title: Efficacy Study of CHG Regimen vs Decitabine to Treat Higher-risk MDS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiao Li (Other)
Responsible Party: Sponsor-Investigator, Xiao Li, Doctor, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHG-DAC 001; SHDC12010202 (Other Grant/Funding Number: Shanghai Shenkang Center for hospital development)
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: myelodysplastic syndromes; Decitabine; homoharringtonine; cytarabine; G-CSF
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Drug Therapy; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHG regimen (Experimental): one course of CHG regimen (low-dose cytarabine, homoharringtonine and G-CSF priming)
  Interventions: Drug: CHG regimen
- Decitabine (Active Comparator): one course of Decitabine (5-aza-deoxycytidine,Dacogen)
  Interventions: Drug: 5-aza-deoxycytidine

INTERVENTIONS:
Drug: CHG regimen — cytarabine (25mg/d, days1-14) and homoharringtonine (1mg/d, days1-14) by intravenous continuous infusion, G-CSF (300 μg/d) by subcutaneous injection from day 0 until neutrophil count recovery to 2.0× 109/L.
  Other Names: Low dose chemotherapy
  Arms: CHG regimen
Drug: 5-aza-deoxycytidine — Decitabine (5-aza-deoxycytidine)for injection, 20mg/m2/day, IV (in the vein) on days 1-5 of each 28 day cycle, Number of Cycles: 2.
  Other Names: Dacogen
  Arms: Decitabine

SUMMARY:
The purpose of this study is to compare the efficacy of CHG regimen (low-dose cytarabine, homoharringtonine with G-CSF priming) to decitabine in the treatment of higher-risk myelodysplastic syndromes(MDS).

DETAILED DESCRIPTION:
Patients with higher-risk myelodysplastic syndrome (MDS) have a survival rate of 0.4 to 1.2 years as well as a high risk of their disease progressing to acute myeloid leukemia (AML). The only treatment with a curative potential is allogeneic stem cell transplantation. However, in the majority of patients, this treatment is not applicable, mainly due to the age of the recipients and comorbid conditions. Low-dose chemotherapy CHG regimen (low-dose cytarabine, homoharringtonine with G-CSF priming)has been used to treat higher-risk MDS in China and achieve high response rate. Hypomethylating agents 5-aza-2'-deoxycytidine (decitabine) is nucleoside analogs that covalently bind to the DNA methyltransferases, irreversibly inhibiting their function, leading to the progressive loss of methylation and reversal of gene silencing. The purpose of this study is to compare the efficacy and safety of CHG regimen to Decitabine in higher-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

* Age rang from 16 to 80 years;
* diagnosis of higher-risk MDS (with≥ 5% blast in bone marrow);
* a performance status of 0-3 according to the Eastern Cooperative Oncology Group (ECOG);
* no evidence of severe concurrent cardiac, pulmonary, neurologic, or metabolic diseases;
* adequate hepatic (serum bilirubin level <2×upper normal limit) and renal (serum creatinine <2×upper normal limit) function tests.

Exclusion Criteria:

* Female with pregnancy;
* a performance of 4-5 according to ECOG score;
* HIV positive;
* uncontrolled severe fungal infection or tuberculosis;
* with other progressive malignant diseases.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | four weeks after one course of CHG or two courses of Decitabine

SECONDARY OUTCOMES:
overall survival | two years
overall remission rate | four weeks after one course of CHG or two courses of Decitabine
disease free survival | two years
hematology toxicities | within the first 4 weeks after CHG or Decitabine regimen
non-hematologic toxicities | within the first 4 weeks after CHG or Decitabine

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Li, Doctor, Study Chair — Shanghai 6th People's Hospital; Lingyun Wu, Doctor, Study Director — Shanghai 6th People's Hospital; Chunkang Chang, Doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality, China